CLINICAL TRIAL: NCT05419232
Title: RADx Up Safe Return to Schools: Strategies to Increase Vaccine Uptake
Brief Title: COVID-19 Vaccine Uptake Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202204166
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Vaccination Refusal; COVID-19
MeSH Terms: conditions — Vaccination Refusal; COVID-19 | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Message Service (SMS) with an associated link to a multi-media website (Active Comparator): The participant will receive a SMS with a brief message containing the following: (1) statement encouraging them to get vaccinated and (2) a link to a multi-media page with videos and additional resources encouraging individuals to be vaccinated. The multi-media website will be housed in the Safe Return To School website and updated by a designated study team members. This page will include the following COVID-19-related resources: publicly available vaccine promotion videos, videos consisting of community members discussing vaccine topics, resources regarding local vaccine sites, and links to additional literature resources.
  Interventions: Other: Short Message Service (SMS) + Website Link Strategy
- Phone Call with Peer (Active Comparator): The participant's peer will be a study team member who has the same or similar racial demographic as the participant. All team members conducting the peer phone calls will be trained in motivational interviewing. The participant will be called by their peer via zoom or phone. Motivational interviewing techniques will be utilized with the participant to promote vaccine uptake. The team member will use a facilitator guide throughout the peer intervention.
  Interventions: Other: Phone Call with Peer Strategy

INTERVENTIONS:
Other: Short Message Service (SMS) + Website Link Strategy — The intervention we are evaluating is the effectiveness of a participant receiving a SMS + Website Link as a vaccine uptake strategy
  Arms: Short Message Service (SMS) with an associated link to a multi-media website
Other: Phone Call with Peer Strategy — The intervention we are evaluating is the effectiveness of a participant having a phone call with a peer as a vaccine uptake strategy
  Arms: Phone Call with Peer

SUMMARY:
The goal of this study is to assess the best COVID-19 vaccine uptake strategy among students, staff and household members that have not been vaccinated.

There is a multitude of recommendations present that highlight different vaccination strategy; however, it is still unclear which strategy is best to increase COVID-19 vaccination rates. We will compare the effectiveness and acceptance of two different communication strategies among unvaccinated students, staff, and their household members.

DETAILED DESCRIPTION:
A sequential multiple assignment randomized trial (SMART) will be conducted to assess two strategies to increase COVID-19 vaccine uptake. The two strategies that will be assessed are a text message with a link to an information website and peer-based motivational interview. If individuals do not seek vaccination after the first intervention, they will again be randomized into the same two interventions. This will allow for testing of both interventions as well as understanding if the use of a more intense intervention (two 'doses') is optimal for vaccine uptake.

In addition, SARS-CoV-2 saliva-based testing will be conducted among students, staff, and household members from the summer of 2022 through the first semester of the 2022-2023 school year. As the pandemic is in its third year, the use of testing among students, staff, and their household members will be assessed Individuals are eligible to be tested multiple times and the testing will occur along different timelines.

ELIGIBILITY:
Inclusion Criteria:

1. Is not up to date with their COVID-19 vaccinations per CDC guidelines
2. is considered eligible by the CDC at the time of enrollment to receive a COVID-19 vaccine
3. is a staff, student, or household member of staff or student of one of the participating school districts OR a resident of St. Louis City or St. Louis County

Exclusion Criteria:

1. Is currently up to date with their COVID-19 vaccinations per CDC guidelines
2. ineligible to receive any COVID-19 vaccine due to medical history or age
3. is not a staff or student, or household member of staff or student of one of the participating school districts AND is not a resident of St. Louis City or St. Louis County
4. participant (or their parents/LAR) do not provide consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Ferguson-Florissant School District, Hazelwood, Missouri
  - Jennings School District, Jennings, Missouri
  - Pattonville School District, Saint Ann, Missouri
  - St. Louis Language Immersion School, St Louis, Missouri
  - Ritenour School District, St Louis, Missouri
  - Normandy Schools Collaborative, St Louis, Missouri
  - Maplewood Richmond Heights School District, St Louis, Missouri
  - University City School District, University City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention. COVID-19; 2022, https://www.cdc.gov/coronavirus/2019-ncov/index.html. Accessed March 1, 2022.
- [Background] Centers for Disease Control and Prevention. COVID-19 Mortality Overview. 2022; https://www.cdc.gov/nchs/covid19/mortality-overview.htm. Accessed March 1, 2022
- [Background] Centers for Disease Control and Prevention. COVID-19; 2022, https://www.cdc.gov/mmwr/volumes/71/wr/mm7101a4.htm#:~:text=COVID%2D19%20vaccines%20are%20highly,death%20(0.0033%25)%20were%20rare., Accessed March 1, 2022
- [Background] Milkman KL, Patel MS, Gandhi L, Graci HN, Gromet DM, Ho H, Kay JS, Lee TW, Akinola M, Beshears J, Bogard JE, Buttenheim A, Chabris CF, Chapman GB, Choi JJ, Dai H, Fox CR, Goren A, Hilchey MD, Hmurovic J, John LK, Karlan D, Kim M, Laibson D, Lamberton C, Madrian BC, Meyer MN, Modanu M, Nam J, Rogers T, Rondina R, Saccardo S, Shermohammed M, Soman D, Sparks J, Warren C, Weber M, Berman R, Evans CN, Snider CK, Tsukayama E, Van den Bulte C, Volpp KG, Duckworth AL. A megastudy of text-based nudges encouraging patients to get vaccinated at an upcoming doctor's appointment. Proc Natl Acad Sci U S A. 2021 May 18;118(20):e2101165118. doi: 10.1073/pnas.2101165118. PMID 33926993
- [Background] Humiston SG, Bennett NM, Long C, Eberly S, Arvelo L, Stankaitis J, Szilagyi PG. Increasing inner-city adult influenza vaccination rates: a randomized controlled trial. Public Health Rep. 2011 Jul-Aug;126 Suppl 2(Suppl 2):39-47. doi: 10.1177/00333549111260S206. PMID 21812168
- [Background] Centers for Disease Control and Prevention. Immunization Strategies for Healthcare Practices and Providers. 2021; https://www.cdc.gov/vaccines/pubs/pinkbook/strat.html . Accessed April 11, 2022
- [Background] Morales-Campos DY, Flores BE, Donovan E, Burdick S, Parra-Medina D, Kahn JA. A qualitative descriptive study of providers' perspectives on human papillomavirus vaccine administration among Latino/a adolescents in South Texas clinics: barriers and facilitators. BMC Public Health. 2022 Mar 5;22(1):443. doi: 10.1186/s12889-022-12837-2. PMID 35248000
- [Background] Shen SC, Dubey V. Addressing vaccine hesitancy: Clinical guidance for primary care physicians working with parents. Can Fam Physician. 2019 Mar;65(3):175-181. PMID 30867173
- [Background] Mehrotra ML, Petersen ML, Geng EH. Understanding HIV Program Effects: A Structural Approach to Context Using the Transportability Framework. J Acquir Immune Defic Syndr. 2019 Dec;82 Suppl 3(Suppl 3):S199-S205. doi: 10.1097/QAI.0000000000002202. PMID 31764255
- [Background] Pearl, J., and E. Bareinboim. External Validity: From Do-Calculus to Transportability Across Populations. Statistical Science. 2014; 29:579-595
- [Background] Dai H, Saccardo S, Han MA, Roh L, Raja N, Vangala S, Modi H, Pandya S, Sloyan M, Croymans DM. Behavioural nudges increase COVID-19 vaccinations. Nature. 2021 Sep;597(7876):404-409. doi: 10.1038/s41586-021-03843-2. Epub 2021 Aug 2. PMID 34340242
- [Background] Almirall D, Nahum-Shani I, Sherwood NE, Murphy SA. Introduction to SMART designs for the development of adaptive interventions: with application to weight loss research. Transl Behav Med. 2014 Sep;4(3):260-74. doi: 10.1007/s13142-014-0265-0. PMID 25264466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited from previous COVID-19 testing studies. Individuals were eligible for the study if they were an employee, student, or a family member of a student or employees from nine school districts and charter schools in St. Louis or if they were a resident of St. Louis City or County and were completely unvaccinated for COVID-19. Eligibility expanded to include individuals that were not up to date for their COVID-19 vaccine.
Pre-assignment Details: 1558 families were called for recruitment, 666 families were screened, 262 individuals were consented, 251 participants received first randomization
Groups:
- Group 1: Call + Call: Participants were randomized to Call at timepoint one and Call at timepoint two
- Group 2: Call + Text: Participants were randomized to Call at timepoint one and Text at timepoint two.
- Group 3: Text + Call: Participants were randomized to Text at timepoint one and Call at timepoint two.
- Group 4: Text + Text: Participants were randomized to Text at timepoint one and Text at timepoint two.
- Group 5: Call Only: Participants were randomized to Call at timepoint one and did not receive a randomization at timepoint two due to reaching the primary endpoint of vaccination, were lost to follow-up, or the participant withdrew.
- Group 6: Text Only: Participants were randomized to Text at timepoint one and did not receive a randomization at timepoint two due to reaching the primary endpoint of vaccination, were lost to follow-up, or the participant withdrew.
Period: Overall Study
Arm/Group | Group 1: Call + Call | Group 2: Call + Text | Group 3: Text + Call | Group 4: Text + Text | Group 5: Call Only | Group 6: Text Only
Started | 56 | 63 | 52 | 71 | 6 | 3
Completed | 53 | 63 | 52 | 71 | 2 | 0
Not Completed | 3 | 0 | 0 | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Call + Call | Group 2: Call + Text | Group 3: Text + Call | Group 4: Text + Text | Group 5: Call Only | Group 6: Text Only | Total
Number analyzed (Participants) | 56 | 63 | 52 | 71 | 6 | 3 | 251
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 38 [14 to 47] | 21 [13 to 43] | 39 [14 to 49] | 30 [13 to 44] | 47 [18.75 to 53.5] | 35 [34 to 51] | 35 [14 to 46]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 44 | 35 | 35 | 47 | 6 | 2 | 169
  Male | 12 | 28 | 17 | 23 | 0 | 1 | 81
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 0 | 3 | 0 | 0 | 11
  Not Hispanic or Latino | 52 | 54 | 50 | 68 | 6 | 3 | 233
  Unknown or Not Reported | 1 | 4 | 2 | 0 | 0 | 0 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 39 | 31 | 29 | 33 | 1 | 2 | 135
  White | 14 | 23 | 18 | 32 | 4 | 1 | 92
  More than one race | 2 | 0 | 2 | 1 | 1 | 0 | 6
  Unknown or Not Reported | 1 | 9 | 3 | 4 | 0 | 0 | 17
Received COVID-19 Vaccine [Count of Participants; unit: Participants] — Participant's COVID-19 Vaccine Status at Enrollment
  Participants
    Yes | 24 | 28 | 20 | 37 | 4 | 1 | 114
    No | 32 | 35 | 32 | 34 | 2 | 2 | 137

OUTCOME MEASURES:

1. Primary Outcome: Vaccine Uptake
Description: The primary outcome of this study will be the percentage of individuals who received any COVID-19 vaccination within two weeks of a study intervention. Vaccine uptake will be primarily assessed by verbal confirmation of recent vaccination during a follow-up visit with a study team member.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Call + Call | Group 2: Call + Text | Group 3: Text + Call | Group 4: Text + Text | Group 5: Call Only | Group 6: Text Only
Number analyzed (Participants) | 56 | 63 | 52 | 71 | 6 | 3
Participants | 1 | 3 | 1 | 0 | 2 | 0

2. Secondary Outcome: Vaccinated or Indicated They Would Receive Vaccine
Description: The primary outcome of this study will be the percentage of individuals who received any COVID-19 vaccination or indicated they would receive any COVID-19 vaccination within two weeks of a study intervention. Vaccine uptake will be primarily assessed by verbal confirmation of recent vaccination during a follow-up visit with a study team member.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Call + Call | Group 2: Call + Text | Group 3: Text + Call | Group 4: Text + Text | Group 5: Call Only | Group 6: Text Only
Number analyzed (Participants) | 56 | 63 | 52 | 71 | 6 | 3
Participants | 7 | 7 | 4 | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Group 1: Call + Call | Group 2: Call + Text | Group 3: Text + Call | Group 4: Text + Text | Group 5: Call Only | Group 6: Text Only
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/63 | 0/52 | 0/71 | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/63 | 0/52 | 0/71 | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/56 | 0/63 | 0/52 | 0/71 | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/32/NCT05419232/Prot_SAP_000.pdf